CLINICAL TRIAL: NCT01176669
Title: A Single-Institutional Phase IIa Trial and A Multi-Institutional Phase IIb Trial of Apatinib in Metastatic Triple-Negative Breast Cancer
Brief Title: Study of Apatinib in Metastatic Triple-Negative Breast Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Xichun Hu, Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Fudan BR2010-03
Record Dates: First submitted 2010-07-20; First posted 2010-08-06 (Estimated); Last update posted 2015-09-09 (Estimated); Status verified 2015-09

CONDITIONS: Metastatic Breast Cancer
Keywords: Apatinib; Triple-Negative Breast Cancer; Metastatic Breast Cancer; ER/PR Negative; Her2/Neu Negative
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Apatinib (Experimental)
  Interventions: Drug: Apatinib

INTERVENTIONS:
Drug: Apatinib — Apatinib was administratered at 750 mg/d in Phase IIa. The actual average dose intensity delivered was 525 mg/d due to toxicities. So, in Phase IIb, the starting dose of apatinib will be 500mg/d. Two dose reductions will be allowed to 375 and then 250 mg/d.
  Other Names: Target therapy

SUMMARY:
The hypothesis of this clinical research study is to discover if the study drug apatinib can shrink or slow the growth of pretreated metastatic triple-negative breast cancer.

DETAILED DESCRIPTION:
Apatinib is a tyrosine kinase inhibitor targeting vascular endothelial growth factor receptor (VEGFR), and its anti-angiogenesis effect has been viewed in preclinical tests. The investigators' phase I study has shown that the drug's toxicity is manageable and the maximum tolerable daily dose is 850 mg. The hypothesis of this clinical research study is to discover if the study drug apatinib can shrink or slow the growth of triple-negative breast cancer. The safety of apatinib will also be studied. Patients physical state, symptoms, changes in the size of the tumor, and laboratory findings obtained while on-study will help the research team decide if apatinib is safe and effective in pretreated metastatic triple-negative breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 and ≤ 70 years of age.
* ECOG performance status of 0-1.
* Women diagnosed with triple negative breast cancer (breast cancer is estrogen receptor negative (ER-), progesterone receptor negative (PgR-) and human epidermal growth factor receptor negative (HER2-). HER2- is defined as 0 or 1+ staining on immunohistochemistry or FISH/CISH negative for gene amplification.
* Metastatic breast cancer, confirmed by histological analysis.
* Have failed for at least one chemotherapy regimen, but at most three regimens(including adjuvant and neo-adjuvant setting).
* Duration from the last therapy (chemotherapy, radiotherapy, target therapy and operation) is more than 4 weeks (Duration for nitroso or mitomycin is 6 weeks).
* Have at least one extracranial measurable site of disease according to RECIST 1.1 criteria that has not been previously irradiated. If the patient has had previous radiation to the marker lesion(s), there must be evidence of disease progression since the radiation.
* Life expectancy of more than 3 months.
* If the patients have brain or meninges metastases, the lesions must have been controlled at least 8 weeks.
* Adequate hepatic, renal, heart, and hematologic functions (hemoglobin ≥ 9.0g/dl, neutrophils ≥ 1.5×10^9/L, platelets ≥ 80×10^9/L , ALT ≤ 2.5 x upper limit of normal (ULN), AST ≤ 2.5 x ULN, serum bilirubin ≤ 1.5 x ULN, serum creatine ≤ 1.5 x ULN, creatinine clearance rate ≥ 50ml/min, PT, APTT, TT, Fbg normal).
* Written informed consent prior to study specific screening procedures, with the understanding that the patient has the right to withdraw from the study at any time without prejudice.

Exclusion Criteria:

* Pregnant or lactating women.
* Less than 4 weeks from the last clinical trial.
* Have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study such as: Congestive heart failure: New York Heart Association Class III/IV, Unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction within 6 months of start of study drug, serious uncontrolled cardiac arrhythmia or any other clinically significant cardiac disease.
* Any factors that influence the usage of oral administration.
* Receiving the therapy of thrombolysis or anticoagulation.
* Unhealed wound or bone fracture.
* Urine protein ≥++ and confirmed >1.0 g by the 24h quantity.
* Previous or present history of pulmonary fibrosis,interstitial pneumonia,pneumoconiosis,radiation pneumonitis,drug-related pneumonitis or greatly-impaired pulmonary function.
* Disability of serious uncontrolled intercurrence infection.
* Abuse of alcohol or drugs.
* Have received prior treatment with a VEGFR, PDGFR or s-SRC TKI (Bevacizumab is permitted).
* History of other malignancies except cured basal cell carcinoma of skin and carcinoma in-situ of uterine cervix.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-06; Primary Completion 2014-06 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
DCR(Disease control rate) for IIa | 8 Weeks
PFS(Progression free survival) for IIb | 8 Weeks

SECONDARY OUTCOMES:
PFS(Progression free survival) for IIa | 8 Weeks
OS (Overall survival) | 8 Weeks
ORR (Objective response rate) | 8 Weeks
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 8 weeks
QoL (Quality of life) | 8 Weeks
DCR(Disease control rate) for IIb | 8 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Xichun Hu, Doctorship, Study Chair — Fudan University
Locations (1):
- Fudan University Cancer Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Fan M, Zhang J, Wang Z, Wang B, Zhang Q, Zheng C, Li T, Ni C, Wu Z, Shao Z, Hu X. Phosphorylated VEGFR2 and hypertension: potential biomarkers to indicate VEGF-dependency of advanced breast cancer in anti-angiogenic therapy. Breast Cancer Res Treat. 2014 Jan;143(1):141-51. doi: 10.1007/s10549-013-2793-6. Epub 2013 Dec 1. PMID 24292957